CLINICAL TRIAL: NCT00587626
Title: Proposal to Evaluate the Efficacy of the InterX 5000 in the Treatment of Chronic Neck and Shoulder Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Memorial Chiropractic College (Other); Neuro Resource Group (Industry)
Responsible Party: Linda J. Woodhouse, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NRG
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-06

CONDITIONS: Neck Pain; Shoulder Pain; Cervical Pain
Keywords: neck pain; shoulder pain; cervical pain; chronic; recurrent
MeSH Terms: conditions — Neck Pain; Shoulder Pain; Bronchiolitis Obliterans Syndrome; Recurrence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): InterX treatment plus rehabilitation exercises
  Interventions: Device: InterX 5000 Treatment
- 2 (Placebo Comparator): Inactive InterX treatment plus rehabilitation exercises
  Interventions: Device: Inactive InterX 5000

INTERVENTIONS:
Device: Inactive InterX 5000 — Patients will receive will receive InterX placebo treatment 3 times a week for 4 weeks.
  Arms: 2
Device: InterX 5000 Treatment — Patients will receive will receive InterX treatment 3 times a week for 4 weeks.
  Arms: 1

SUMMARY:
The purpose of the proposed study is to evaluate the efficacy of the InterX 5000 in relieving chronic neck and shoulder pain. This study will focus on the efficacy of treating patients who have functional limitations in activity because of chronic/recurrent neck or shoulder pain.

H1: InterX therapy will have a moderate effect to reduce pain.

H2: Functional gains will be greater in patients receiving InterX therapy compared to those who received placebo treatment.

H3: Chronic neck and shoulder pain is more prevalent in patients who exhibit radiographic evidence of degenerative spondylosis/arthrosis of the cervical spine.

DETAILED DESCRIPTION:
Electrical stimulation modalities of various types have been used as a therapeutic intervention for years in a wide variety of applications. Individuals with neck and shoulder pain represent a significant segment of the pain population seeking relief. However, there is a paucity of data from quality studies published in mainstream peer-reviewed journals supporting the effectiveness of this intervention. No well-designed prospective, randomized, controlled trials investigating the efficacy or effectiveness of this intervention in patients with chronic neck and shoulder pain have been reported. The need for such work is becoming increasingly important considering the progressively greater demands for evidence-based medicine to justify reimbursement for care.

ELIGIBILITY:
Inclusion Criteria:

* chronic or recurrent neck or shoulder pain of at least 3 months duration with or without arm pain
* willing to sign consent for study participation
* able/willing to comply with treatment schedule

Exclusion Criteria:

* clinically significant herniated disc (defined as positive radicular arm pain aggravated by head position change or neural stretch signs from provocative arm movement, this will not exclude patients with any imaged herniation as this is a common finding in all populations)
* spinal fracture
* previous electrical stimulation treatment for this episode
* recent cervical spinal or shoulder surgery or implanted instrumentation/prostheses.
* patients with cardiac pacemaker or spinal cord stimulator, epilepsy, pregnancy, recent (3 months) chemotherapy/radiotherapy, phlebitis, cortisone use (30 days)

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 4 weeks
Neck Disability Index (NDI) | 4 weeks
Medical Outcomes Study Short-Form 36 (SF-36) Health Survey | 4 weeks
Short-Form McGill Questionnaire | 4 weeks
Biomarkers (inflammatory cytokines and SP) | 4 weeks
Functional Impairment Test-Hand, and Neck, Shoulder, Arm (FIT-HaNSA) | 4 weeks
Cervical Range of Motion (CROM) | 4 weeks
Grip strength | 4 weeks
Vibration threshold | 4 weeks
Pain Tolerance and Threshold - Pressure | 4 weeks
Pain Threshold and Tolerance - Current Perception | 4 weeks
Current Perception Threshold | 4 weeks
Neck Walk Index (NWI) | 4 weeks
Muscle Fatigue | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Linda J Woodhouse, PhD, Principal Investigator — McMaster University; John J Triano, DC, PhD, Principal Investigator — Canadian Memorial Chiropractic College; Vickie Galea, PhD, Principal Investigator — McMaster University; H Stephen Injeyan, PhD, DC, Principal Investigator — Canadian Memorial Chiropractic College; Joy MacDermid, PhD, Principal Investigator — McMaster University; Marion McGregor, DC, PhD, Principal Investigator — Canadian Memorial Chiropractic College; Michael Pierrynowski, PhD, Principal Investigator — McMaster University; Richard Ruegg, PhD, DC, Principal Investigator — Canadian Memorial Chiropractic College; Julita A Teodorczyk-Injeyan, PhD, Principal Investigator — Canadian Memorial Chiropractic College
Locations (2):
- Canada (2):
  - McMaster University, Hamilton, Ontario
  - Canadian Memorial Chiropractic College, Toronto, Ontario